CLINICAL TRIAL: NCT03225469
Title: Improving Effect of Reinforced Family Member Education on the Quality of Bowel Preparation for Colonoscopy
Brief Title: Improving Effect of Reinforced Family Assistance on the Quality of Bowel Preparation for Colonoscopy
Acronym: IERFAOBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Zql201706
Record Dates: First submitted 2017-07-15; First posted 2017-07-21 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Bowel Preparation
Keywords: Bowel Preparation; Colonoscopy; Quality; Family Support; Education

STUDY DESIGN:
Intervention Model Description: reinforced family member education group, regular education (control) group
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients and the associated family members know which group they are assigned，while the colonoscopist, information collector are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reinforced family member education group (Experimental): Regular instructions will be given to all patients during the colonoscopy appointment. At least one family member who lives with the patient together will be given instruction at the basis of patent education.
  Interventions: Behavioral: reinforced family member education
- regular education group (No Intervention): Regular instructions will be given to the patients during the colonoscopy appointment. There will be nothing specially for family members.

INTERVENTIONS:
Behavioral: reinforced family member education — Based on regular instructions for patent education, at least one family member who lives with the patient together will be given special instruction.
  Other Names: reinforced family member instruction
  Arms: reinforced family member education group

SUMMARY:
Enhanced instructions such as re-education by telephone or short message which increase the patient adherence eventually improve the quality of bowel preparation significantly. However, the effect of family assistance which plays an essential role on compliance of patient with treatment on bowel preparation is unknown. The investigators hypothesized that reinforced education giving family members of outpatients will enhance family support to patients for colonoscopy, and consequently improve the quality of bowel preparation.

Therefore, the investigators designed protocols to reinforce family member education by verbal (face to face or telephone) and written methods. The aim of this study is to evaluate the effect of reinforced family member education on patient compliance and the quality of bowel preparation for colonoscopy. In addition，the rate of side effects happening, the subjective feelings of bowel preparation, the outcomes of colonoscopy ,and the independent risk factors will be also assessed.

DETAILED DESCRIPTION:
Adequate bowel preparation is essential for optimal examination of the colorectal mucosa during colonoscopy. However, approximately 10%-30% bowel preparation is inadequate, leading to significantly decrease diagnostic accuracy and surveillance intervals, increase the procedural difficulties, and even increase the procedure-related complications. As reported, enhanced instructions such as re-education by telephone or short message which increase the patient adherence eventually improve the quality of bowel preparation significantly. However, the effect of family assistance which plays an essential role on compliance of patient with treatment on bowel preparation is unknown. The investigators hypothesized that reinforced education giving family members of outpatients will enhance family support to patients for colonoscopy, and consequently improve the quality of bowel preparation.

Therefore, the investigators designed protocols to reinforce family member education by verbal (face to face or telephone) and written methods. The aim of this study is to evaluate the effect of reinforced family member education on patient compliance and the quality of bowel preparation for colonoscopy. In addition，the rate of side effects happening, the subjective feelings of bowel preparation, the outcomes of colonoscopy ,and the independent risk factors will be also assessed.

This is a prospective, endoscopist-blinded, randomized, controlled study.

1. Patients, Arm Description, Education and Blinding. Consecutive individuals over 18 years, who will be scheduled for undergoing colonoscopy between September and December 2017 at the Endoscopy Center of Wuxi people's Hospital in China and are not accord with the exclusion criteria will be enrolled in the study. After signature of informed consent, Patients will be consecutively randomized to either the reinforced family member education (RFME) or regular education (control) group at the time of colonoscopy appointments by opening a sealed opaque envelope. Regular instructions will be given to all patients during the colonoscopy appointment by one experienced endoscopy nurse. For RFME group, at least one family member who lives with the patient together will be given instruction at the basis of patent education. The information of group assignments will be keep from colonoscopists and other investigators at any time.
2. Bowel preparation. Two kinds of purgatives, magnesium sulphate and polyethylene glycol electrolyte powder (PEG-ELP), are available in our endoscopy center, and the type will be prescribed by physician based on the conditions of the patient.
3. Data collection and Definitions. On the day of colonoscopy, the patients will be asked to arrive at the Endoscopy Center 1 h before the procedure. The baseline data, clinical data and related data of the enrolled patients will be collected 1 h before the colonosc0py.
4. Colonoscopy. All colonoscopy will be carried out between 13:30 and 16:30 by 5 five experienced endoscopists. The Boston Bowel Preparation Scale (BBPS) scoring system will be employed for the assessment of the quality of bowel preparation. The endoscopists will be asked to give the BBPS score immediately after the colonoscopy, and the findings of the colonoscopy, the cecal intubation, the insertion time, the withdrawal time and the incomplete examination cases not for poor bowel preparation will be recorded simultaneously.
5. Statistical analysis. A total of 276 patients in each group will be required to obtain statistical significance for the primary outcome. Baseline characteristics, primary and secondary outcomes will be evaluated by intention-to-treat (ITT) analysis. To assess independent risk factors associated with inadequate bowel preparation, multivariate analysis will be conducted using the score of bowel preparation quality (BBPS <5) with a P value of ≤ 0.10 in the univariate analysis. All analyses will be carried out with SPSS software V.20.0 (SPSS Inc., Chicago, IL, USA). A P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals scheduled for undergoing colonoscopy at the Endoscopy Center of Wuxi people's Hospital in China
2. Greater than the age of 18
3. Individuals living with other family members
4. Outpatients

Exclusion criteria:

1. History of colorectal surgery
2. Suspected or known digestive tract obstruction, stricture, or perforation
3. Serious status of illness, such as severe renal failure whose creatinine clearance<30 ml/min, New York Heart Association grade III or grade IV congestive heart failure, or hemodynamic instability, etc.
4. Incapable of completing bowel preparation，such as dysphagia, allergy to purgatives, or impaired mental status, etc.
5. Pregnancy or breastfeeding
6. Incomplete colonoscopy due to causes except poor bowel preparation
7. Unable to give informed consent
8. Have participated in the study before.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2017-08-15 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
The qualified rate of bowel preparation | 5 months
  The score of Boston Bowel Preparation Scale = > 2 points for each region or = > 5 for the total colon will be considered as adequate bowel preparation to corresponding intestinal segments or total colon.

SECONDARY OUTCOMES:
Patient compliances | 2 days
  Compliance of dietary restrictions, integrity of purgatives ingestion, and water intake, are scored on a three-point scale based on a previous report with a little improvement, as follow：the estimated percentage of fulfilled instructions, high = > 70% getting 3point, moderate = 40% - 70% getting 2points, and low = <40% getting 1point.
The level of family assistance | 2 days
  The level of family assistance is also scored on the three-point scale, = > 70% is defined as that the family member pay much attention to the colonoscopy, actively encourage, assist and supervise the patient to complete dietary preparation and bowel preparation according to the instruction. And 40% - 70% is that some certain extent supervision and reminders are provided by the family member but not actively, While = <40% is that the family member only know this examination, and very little encouragement and supervision are provided, or even worse.
The subjective feelings of bowel preparation | 2 days
  The subjective feelings include sleep quality, anxiety levels, and willingness to repeat bowel preparation if necessary.
The rate of cecal intubation | 6 months.
  Proportion of successful cecal intubation individuals in total
The polyp detection rates | 6 months.
  Proportion of polyp detection individuals in total
The insertion and withdrawal time. | 1 day
  The time of insertion and withdrawal during colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhan, senior, Study Director — Wuxi People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided